CLINICAL TRIAL: NCT06121349
Title: The Wearing-off Effect of Anti-CD20 Therapies in Patients With Multiple Sclerosis
Brief Title: WOE of Anti-CD20 Therapies
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157AUS22
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis
Keywords: NIS; Anti-CD20 Therapies; Multiple Sclerosis; OCR; Ocrevus; OMB; KESIMPTA
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab; ofatumumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (2):
- OCR: Patients under treatment with Ocrelizumab (OCR) for at least 1 year prior to study start.
  Interventions: Drug: ocrelizumab
- OMB: Patients under treatment with ofatumumab (OMB) for at least 6 months prior to study start
  Interventions: Drug: ofatumumab

INTERVENTIONS:
Drug: ocrelizumab — infusion therapy administered every six months
  Other Names: Ocrevus
  Groups: OCR
Drug: ofatumumab — self-injectable every month
  Other Names: KESIMPTA
  Groups: OMB

SUMMARY:
The nature, intensity, and prevalence of this wearing-off effect remain poorly understood. To our knowledge, there is no consensus in the literature on what symptoms constitute a wearing-off effect, nor is there a single validated scale that measures wearing-off effect. The current study will explore the wearing-off effect associated with OCR and OMB, using a variety of validated scales assessing MS symptoms (i.e., fatigue, mobility, pain, depression, cognition), as well as some global questions on wearing-off. In addition, impact of worsening of MS symptoms on patients' health-related quality of life (HRQoL) and their work productivity will be assessed using relevant MS-specific validated scales

DETAILED DESCRIPTION:
This will be a non-interventional, primary data collection study in patients with MS treated with an established anti-CD20 treatment regimen (OCR or OMB) in the United States. Patients who satisfy the inclusion criteria and consent to participate in the study will be surveyed at four timepoints at the beginning and the end of OCR or OMB treatment cycles according to the following assessment schedule:

* Assessment 1. 0-10 days before 1st dose post-enrollment (index dose)
* Assessment 2: 5-14 days after index dose
* Assessment 3: 0-10 days before 2nd dose post-enrollment (follow-up dose)
* Assessment 4: 5-14 days after follow-up dose dose

ELIGIBILITY:
Inclusion Criteria:

OCR sample:

* Self-reported diagnosis of RMS, SPMS or CIS
* ≥21 years old at the time of initial contact
* Under treatment with OCR at the time of initial contact
* Have been on OCR for ≥ 1 year at the time of initial contact (i.e., prevalent users)
* Able to answer the questionnaires in English

OMB sample

* Self-reported diagnosis of RMS, SPMS or CIS
* ≥21 years old at the time of initial contact
* Under treatment with OMB at the time of initial contact
* Have been on OMB for ≥6 months at the time of initial contact (i.e., prevalent users)
* Able to answer the questionnaires in English

Exclusion Criteria:

OCR sample:

* Currently participating in a clinical trial involving MS drugs
* Last Ocrevus infusion was less than 3 months back

OMB sample:

Currently participating in a clinical trial involving MS drugs

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with MS who are taking ofatumumab or ocrelizumab
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who experience wearing-off effect | Up to 10 days before index dose (first dose) post enrollment, from 5 to 14 days after index dose, up to 10 days before second dose post enrollment, from 5 to 14 days after second dose.
  The wearing-off effect questionnaire for this study was modified from a pre-existing tool designed by (Toorop, et al., 2022) such that it is now suitable to assess wearing-off in patients on either infusible or self-injectable disease modifying therapies (DMTs) with different dosing intervals. There is no numeric rating scale (NRS) associated with this endpoint.
Proportion of patients with worsening ≥1 category for PROMIS physical health NRS | Up to 10 days before index dose (first dose) post enrollment, from 5 to 14 days after index dose, up to 10 days before second dose post enrollment, from 5 to 14 days after second dose.
  The PROMIS Global-10 is a publicly available global health assessment tool that allows measurements of symptoms, functioning, and healthcare-related quality of life (HRQoL) for a wide variety of chronic diseases and conditions. PROMIS physical health is measured using the item 3 from the PROMIS Global-10. Scale for PROMIS physical health a is from 1 (worst) - 5 (best).
Proportion of patients with worsening ≥ 1 category for PROMIS mental health NRS | Up to 10 days before index dose (first dose) post enrollment, from 5 to 14 days after index dose, up to 10 days before second dose post enrollment, from 5 to 14 days after second dose.
  The PROMIS Global-10 is a publicly available global health assessment tool that allows measurements of symptoms, functioning, and healthcare-related quality of life (HRQoL) for a wide variety of chronic diseases and conditions. PROMIS mental health is measured using the item 4 from the PROMIS Global-10. Scale for PROMIS mental health is from 1 (worst) - 5 (best).
Proportion of patients with worsening ≥ 1 category for PROMIS fatigue NRS | Up to 10 days before index dose (first dose) post enrollment, from 5 to 14 days after index dose, up to 10 days before second dose post enrollment, from 5 to 14 days after second dose.
  The PROMIS Global-10 is a publicly available global health assessment tool that allows measurements of symptoms, functioning, and healthcare-related quality of life (HRQoL) for a wide variety of chronic diseases and conditions. PROMIS fatigue is measured using the item 8r from the PROMIS Global-10. Scale for PROMIS fatigue is from 1 (worst) - 5 (best).
Proportion of patients with worsening ≥1 category for PROMIS pain NRS | Up to 10 days before index dose (first dose) post enrollment, from 5 to 14 days after index dose, up to 10 days before second dose post enrollment, from 5 to 14 days after second dose
  The PROMIS Global-10 is a publicly available global health assessment tool that allows measurements of symptoms, functioning, and healthcare-related quality of life (HRQoL) for a wide variety of chronic diseases and conditions. PROMIS pain is measured using the item 7rc from the PROMIS Global-10. Scale for PROMIS fatigue is from 0 (worst) - 10 (best).
Median score change for the physical health, mental health, fatigue and pain domains of PROMIS NRS | Up to 10 days before index dose (first dose) post enrollment, from 5 to 14 days after index dose, up to 10 days before second dose post enrollment, from 5 to 14 days after second dose.
  PROMIS is a publicly available system of highly reliable, precise measures of patient-reported health status relevant to a variety of chronic conditions including MS.
  Mean score change for PROMIS physical health, mental health fatigue and pain NRS to be provided.
Proportion of patients with worsening ≥ 1 category for Neuro-QoL fatigue scale | Up to 10 days before index dose (first dose) post enrollment, from 5 to 14 days after index dose, up to 10 days before second dose post enrollment, from 5 to 14 days after second dose.
  Neuro-QoL is a publicly available set of self-report measures that assesses the HRQoL of adults and children with neurological disorders. Neuro-QoL is comprised of item banks and scales that evaluate symptoms, concerns, and issues that are relevant across disorders along with instruments that assess areas most relevant for specific patient populations. The Neuro-Qol fatigue scale is an eight-item short form with a scale ranging from 29.5 (best) - 74.1 (worst).
Median score change for Neuro-QoL fatigue scale | Up to 10 days before index dose (first dose) post enrollment, from 5 to 14 days after index dose, up to 10 days before second dose post enrollment, from 5 to 14 days after second dose.
  Neuro-QoL is a publicly available set of self-report measures that assesses the HRQoL of adults and children with neurological disorders. Neuro-QoL is comprised of item banks and scales that evaluate symptoms, concerns, and issues that are relevant across disorders along with instruments that assess areas most relevant for specific patient populations. The Neuro-Qol fatigue scale is an eight-item short form with a scale ranging from 29.5 (best) - 74.1 (worst).
Proportion of patients with worsening ≥ Minimal Clinically Important Difference (MCID) for Fatigue Severity Scale (FSS) | Up to 10 days before index dose (first dose) post enrollment, from 5 to 14 days after index dose, up to 10 days before second dose post enrollment, from 5 to 14 days after second dose.
  The FSS is a publicly available, self-report, nine-item instrument designed to assess fatigue as a symptom of a variety of different chronic conditions and disorders. Answers are scored on a seven-point scale where 1 corresponds to strongly disagreeing and 7 corresponds to strongly agreeing. Scale for FSS is from 9 (best) - 63 (worst), or 1 (best) - 7 (worst) if the mean of all the scores is reported. The MCID for the mean FSS score is in the 0.5-1.1 range based on (Robinson, et al., 2009)
Mean score change for Fatigue Severity Scale (FSS) | Up to 10 days before index dose (first dose) post enrollment, from 5 to 14 days after index dose, up to 10 days before second dose post enrollment, from 5 to 14 days after second dose.
  The FSS is a publicly available, self-report, nine-item instrument designed to assess fatigue as a symptom of a variety of different chronic conditions and disorders. Answers are scored on a seven-point scale where 1 corresponds to strongly disagreeing and 7 corresponds to strongly agreeing. Scale for FSS is from 9 (best) - 63 (worst), or 1 (best) - 7 (worst) if the mean of all the scores is reported. The MCID for the mean FSS score is in the 0.5-1.1 range based on (Robinson, et al., 2009)
Proportion of patients with worsening ≥ significant individual difference (SID) for Neuro-QoL mobility scale | Up to 10 days before index dose (first dose) post enrollment, from 5 to 14 days after index dose, up to 10 days before second dose post enrollment, from 5 to 14 days after second dose.
  Neuro-QoL is a publicly available set of self-report measures that assesses the HRQoL of adults and children with neurological disorders. Neuro-QoL is comprised of item banks and scales that evaluate symptoms, concerns, and issues that are relevant across disorders along with instruments that assess areas most relevant for specific patient populations. The Neuro-Qol mobility scale is an eight-item short form with a scale ranging from 16.5 (worst) - 58.6 (best).
Proportion of patients with worsening ≥ SID for Neuro-QoL depression scale | Up to 10 days before index dose (first dose) post enrollment, from 5 to 14 days after index dose, up to 10 days before second dose post enrollment, from 5 to 14 days after second dose.
  Neuro-QoL is a publicly available set of self-report measures that assesses the HRQoL of adults and children with neurological disorders. Neuro-QoL is comprised of item banks and scales that evaluate symptoms, concerns, and issues that are relevant across disorders along with instruments that assess areas most relevant for specific patient populations. The Neuro-Qol depression scale is an eight-item short form with a scale ranging from 36.9 (best) - 75.0 (worst).
Proportion of patients with worsening ≥ SID for Neuro-QoL cognition scale | Up to 10 days before index dose (first dose) post enrollment, from 5 to 14 days after index dose, up to 10 days before second dose post enrollment, from 5 to 14 days after second dose.
  Neuro-QoL is a publicly available set of self-report measures that assesses the HRQoL of adults and children with neurological disorders. Neuro-QoL is comprised of item banks and scales that evaluate symptoms, concerns, and issues that are relevant across disorders along with instruments that assess areas most relevant for specific patient populations. The Neuro-Qol cognition scale is an eight-item short form with a scale ranging from 17.3 (worst) - 64.2 (best).
Mean score change for Neuro-QoL mobility, depression and cognition domains | Up to 10 days before index dose (first dose) post enrollment, from 5 to 14 days after index dose, up to 10 days before second dose post enrollment, from 5 to 14 days after second dose.
  Neuro-QoL is a publicly available set of self-report measures that assesses the HRQoL of adults and children with neurological disorders. Neuro-QoL is comprised of item banks and scales that evaluate symptoms, concerns, and issues that are relevant across disorders along with instruments that assess areas most relevant for specific patient populations.

SECONDARY OUTCOMES:
Mean score change for both domains (physical impact and psychological impact) of Multiple Sclerosis Impact Scale (MSIS-29) | Up to 10 days before index dose (first dose) post enrollment, from 5 to 14 days after index dose, up to 10 days before second dose post enrollment, from 5 to 14 days after second dose.
  The MSIS-29 questionnaire evaluates the influence of MS-related symptoms on physical and psychological functioning in daily life and contains 29 questions, of which 20 address the physical impact component and nine assess the psychological impact. Physical and psychological scale scores are generated by summing individual items and then transformed to a 0 (best) -100 (worst) scale.
Proportion of patients with worsening ≥ MCID for the MSIS-29 | Up to 10 days before index dose (first dose) post enrollment, from 5 to 14 days after index dose, up to 10 days before second dose post enrollment, from 5 to 14 days after second dose.
  The MSIS-29 questionnaire evaluates the The MSIS-29 questionnaire evaluates the influence of MS-related symptoms on physical and psychological functioning in daily life and contains 29 questions, of which 20 address the physical impact component and nine assess the psychological impact. Physical and psychological scale scores are generated by summing individual items and then transformed to a 0 (best) -100 (worst) scale. The MCID for the physical impact score (6.8) and psychological impact score (7.4) are based on the work from (Greene, et al., 2023).
Mean score change for each of the 4 domains of the Work Productivity and Activity Impairment Questionnaire for MS (WPAI:MS) | Up to 10 days before index dose (first dose) post enrollment, from 5 to 14 days after index dose, up to 10 days before second dose post enrollment, from 5 to 14 days after second dose.
  The Work Productivity and Activity Impairment: MS (WPAI:MS) questionnaire is a well validated instrument measuring the effect of MS on work productivity and regular activities during the past seven days. The questions are computed according to specific calculation rules and have four scores: (1) percentage work time missed due to health (absenteeism); (2) percentage impairment at work due to health (presenteeism); (3) percentage overall work productivity loss due to MS; and (4) percentage daily activity impairment outside of work due to MS. Scale for each of the 4 domains is 0% (best) - 100% (worst).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No